CLINICAL TRIAL: NCT03899987
Title: Randomized Phase 2 Study: Neoadjuvant Conditioning of Prostate Cancer Tumor Microenvironment Using a Novel Chemokine-Modulating Regimen
Brief Title: Aspirin and Rintatolimod With or Without Interferon-alpha 2b in Treating Patients With Prostate Cancer Before Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 77318; NCI-2019-01192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 77318 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-03-15; First posted 2019-04-02 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Aspirin; Introns; Interferon alpha-2; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm I (EC aspirin, interferon alpha, rintatolimod, surgery) (Experimental): Patients receive aspirin PO BID on days -7 to 7. Patients also receive recombinant interferon alfa-2b IV over 20 minutes and rintatolimod IV over 2 hours on days 1-3 and 8-10 in the absence of disease progression or unacceptable toxicity. Patients then undergo radical prostatectomy on or between day 17-24..
  Interventions: Drug: EC Aspirin; Procedure: Radical Prostatectomy; Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod
- Arm II (EC aspirin, rintatolimod, surgery) (Experimental): Patients receive aspirin PO BID on days -7 to 7 and rintatolimod IV over 2 hours on days 1-3,and 8-10 in the absence of disease progression or unacceptable toxicity. Patients then undergo radical prostatectomy on or between day 17-24.
  Interventions: Drug: EC Aspirin; Procedure: Radical Prostatectomy; Drug: Rintatolimod
- Arm III (radical prostatectomy) (Active Comparator): Patients undergo radical prostatectomy about 4 weeks after enrollment.
  Interventions: Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: EC Aspirin — Given PO
  Other Names: Acetylsalicylic Acid; ASA; Aspergum; aspirin; Ecotrin; Empirin; Entericin; Extren; Measurin; Enteric-coated aspirin
  Arms: Arm I (EC aspirin, interferon alpha, rintatolimod, surgery); Arm II (EC aspirin, rintatolimod, surgery)
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy
Biological: Recombinant Interferon Alfa-2b — Given IV
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
  Arms: Arm I (EC aspirin, interferon alpha, rintatolimod, surgery)
Drug: Rintatolimod — Given IV
  Other Names: Ampligen; Atvogen
  Arms: Arm I (EC aspirin, interferon alpha, rintatolimod, surgery); Arm II (EC aspirin, rintatolimod, surgery)

SUMMARY:
This phase II trial studies how well enteric-coated (EC) aspirin and rintatolimod with or without interferon-alpha 2b work in treating patients with prostate cancer before surgery. EC Aspirin may help to keep the prostate cancer from coming back. Rintatolimod may stimulate the immune system and interfere with the ability of tumor cells to grow and spread. Interferon-alpha 2b may improve the body's natural response to infections and may slow tumor growth. It is not yet known how well rintatolimod, EC aspirin, and interferon-alpha 2b work in treating patients with prostate cancer undergoing surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the immunomodulatory effectiveness of the combination of rintatolimod and EC aspirin with or without recombinant interferon alfa-2b (interferon [IFN]-alpha), in participants with localized prostate cancer undergoing radical prostatectomy.

SECONDARY OBJECTIVES:

I. Assess the safety and toxicity of the treatment combinations in participants with localized prostate cancer undergoing radical prostatectomy.

II. Assess the antitumor activity between treatment arms.

EXPLORATORY OBJECTIVES:

I. Compare the resected tumor tissue specimen and surrounding tissue samples of both study arms (pre versus [vs] post-chemokine modulatory [CKM] treatment, with vs without CKM, CKM doublet vs CKM triplet) with regards to infiltrating T cell subtypes, effector T cell (Teff)/regulatory T cell (Treg) ratios, CD11b+ myeloid-derived suppressor cell (MDSC); the expression of chemokine receptors and immune checkpoint molecules on immune cells; local expression of Teff-attracting chemokines and Treg/MDSC-favoring chemokines; ribonucleic acid (RNA) signatures of groups of immune-regulatory genes that are modulated by the CKM regimen.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive EC aspirin orally (PO) two times a day (BID) from day -7 to 7 days prior to surgery. Patients also receive recombinant interferon alfa-2b intravenously (IV) over 20 minutes and rintatolimod IV over 2 hours on days 1-3, and 8-10 in the absence of disease progression or unacceptable toxicity. Patients then undergo radical prostatectomy on or between day 17-24.

ARM II: Patients receive EC aspirin PO BID from day -7 to 7 days prior to surgery and rintatolimod IV over 2 hours on days 1-3 and 8-10 in the absence of disease progression or unacceptable toxicity. Patients then undergo radical prostatectomy on or between day 17-24.

ARM III: Patients undergo radical prostatectomy about 4 weeks after enrollment.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, localized prostate adenocarcinoma patients who are planning to have a radical prostatectomy.
* Diagnostic prostate biopsy must have been obtained within 6 months patients who had biopsies at outside facilities may be eligible if tissue availability and adequacy can be confirmed by pathology.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Platelet >= 75,000/uL.
* Hemoglobin >= 9 g/dL.
* Hematocrit >= 27%.
* Absolute neutrophil count (ANC) >= 1500/uL.
* Creatinine < institutional upper limit of normal (ULN) OR creatinine clearance >= 50 mL/min for patients with creatinine levels greater than ULN.
* Total bilirubin =< 1.5 X institutional ULN.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 X institutional ULN.
* Serum amylase and lipase =< 1.5 X institutional ULN.
* Negative hepatitis panel for patients with a history of Hepatitis
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Patients currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 3 weeks after removal from immunosuppressive treatment.
* Patients who received hormonal therapy, 5-alpha reductase inhibitors (such as finasteride, dutasteride), chemotherapy, radiotherapy, major surgery, or biologic therapy within 3 weeks of protocol treatment.
* Patients with active prostatitis.
* Patients with active autoimmune disease or history of transplantation.
* Patients with comorbid medical conditions that render them unfit for surgery.
* Metastatic disease based on preoperative imaging.
* Cardiac risk factors including:

  * Patients experiencing cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent
  * Patients with a New York Heart Association classification of III or IV.
* History of upper and lower gastrointestinal ulceration, upper gastrointestinal bleeding, or perforation within the past 3 years.
* History of bleeding disorders, known lesions at risk for bleeding, or history of recent clinically significant bleed or hemorrhage (<3months).
* Prior allergic reaction or hypersensitivity to aspirin, or other nonsteroidal antiinflammatory drugs (NSAIDs).
* Patients are ineligible if they plan on use of other NSAIDs at any dose during the trial. Patients who agree to stop regular NSAIDs are eligible and no wash out period is required.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator?s opinion deems the participant an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
Count of tumor infiltrating CD8+ lymphocytes | Up to 3 years
  This will be assessed by the increase in the total number of tumor infiltrating CD8+ T cells in the radical prostatectomy specimen (measured as cell density of CD8+ cell by immunohistochemistry), comparing Arm A versus Arm B versus Arm C. Will be natural log transformed prior to analysis. The primary analysis will consist of testing the single degree of freedom planned contrast at alpha = .10 that the 3 treatment means are in the ratio of 3:2:1 (contrast coefficients 3, -2, -1) for groups A, B and C, respectively groups. If this test rejects the null hypothesis of no group differences, will proceed to estimate group means and pairwise differences between groups with 90% confidence intervals. Non-overlapping confidence intervals will serve as evidence of differential treatment effects.

SECONDARY OUTCOMES:
Pathologic response | Up to 3 years
  Spearman rank correlation coefficients will be used to estimate the correlation between CD8+ tumor infiltrate, pathologic response rate and prostate specific antigen (PSA) response.
Number of patients with Surgical margin positivity | Up to 3 years
PSA response | Up to 3 years
  Spearman rank correlation coefficients will be used to estimate the correlation between CD8+ tumor infiltrate, pathologic response rate and PSA response.
Incidence of treatment-related adverse events | Up to 30 days post treatment
  Will be evaluated with National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal S Chatta, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States